CLINICAL TRIAL: NCT04203888
Title: Re-engineering Precision Therapeutics Through N-of-1 Trials
Brief Title: Personalized Trial for Chronic Lower Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Karina Davidson, Senior Vice President of Research, Northwell Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 19-0672
Record Dates: First submitted 2019-11-18; First posted 2019-12-18 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Back Pain Lower Back Chronic
Keywords: N-of-1; Yoga; Massage; Pain; Low Back Pain; Lower Back Pain; Virtual; Swedish Massage; Personalized Trial; Personalized; Feasibility
MeSH Terms: conditions — Pain; Low Back Pain | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: This study utilizes a multiple crossover design to conduct N-of-1 trials in individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Massage (Other): A licensed massage therapist will deliver 60-minute Swedish Massage in the participant's home, 2 times per week with at least 48-hours between massage sessions. Each massage arm will be 2 weeks in length, and consist of 4 total Swedish massages.
  Interventions: Other: Swedish Massage
- Yoga (Other): A certified yoga instructor will deliver 60-minute yoga instruction in the participant's home, 2 times per week with at least 48-hours between yoga session. Yoga sessions will be based on the yoga postures available in the appendix of the December 2005 Annals of Internal Medicine article, "Comparing Yoga, Exercise, and a Self-Care Book for Chronic Low Back Pain" (Sherman KJ et al., 2005). Each yoga arm will be 2 weeks in length, and consist of 4 total yoga sessions.
  Interventions: Other: Yoga
- Usual Care (No Intervention): Participants will be instructed to abstain from any massage or yoga activity, and instructed to treat their chronic lower back pain as they normally would. Each usual care arm will be 2 weeks in length.

INTERVENTIONS:
Other: Swedish Massage — 60-minute Swedish Massage delivered in-home by a licensed massage therapist, 2 times per week with at least 48-hours between massage interventions.
  Arms: Massage
Other: Yoga — 60-minute yoga session delivered in-home by a certified yoga instructor, 2 times per week with at least 48-hours between yoga interventions.Yoga sessions will be based on the yoga postures available in the appendix of the December 2005 Annals of Internal Medicine article, "Comparing Yoga, Exercise, and a Self-Care Book for Chronic Low Back Pain" (Sherman KJ et al., 2005).
  Other Names: Viniyoga
  Arms: Yoga

SUMMARY:
The Personalized Trial of Chronic Lower Back Pain will test the feasibility of employing technology to facilitate remote N-of-1 interventions to research participants with self-identified back pain. Participants will spend 14 weeks alternating between massage, yoga, and usual care methods to treat their back pain, while answering daily questions and wearing an activity tracker. After 14 weeks, participants will have the ability to share their opinions about a Personalized Trials platform. We believe a Personalized Trials platform will be satisfactory to participants and feasible to scale to large randomized controlled trials, and eventually to clinical practice.

DETAILED DESCRIPTION:
The Personalized Trial of Chronic Lower Back Pain will facilitate remote N-of-1 interventions to research participants with self-identified back pain persisting longer than 12 weeks. Participants will be randomized in a multiple crossover design to receive Swedish massage in-home by a commercial wellness service, yoga instruction in-home by a commercial wellness service, and no intervention/usual care. Participants will evaluate their pain intensity, pain interference, fatigue and stress daily through self-reported questionnaires. Online screening and enrollment methods, text-message reminders and questionnaire prompts, and wearable devices will be employed to collect data. At the end of the study, participants will receive a personalized report summarizing their observed data in each treatment period. Participants will evaluate the system usability of Personalized Trials, will debrief their experience with a member of the research team, and will share their overall satisfaction with Personalized Trials.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Fluent in English
* Experiencing symptoms of low back pain for > 12 weeks
* Self-reported pain intensity > 8 on the PROMIS pain intensity scale during screening
* Able to receive massage and yoga interventions (2x/week between 8 am and 10 pm)
* Owns and can regularly access a smartphone capable of receiving text messages
* Owns and can regularly access an e-mail account

Exclusion Criteria:

* Pregnant women
* History of spinal surgery
* Complex back pain (e.g. sciatica, spinal stenosis, or other pre-existing condition)
* Previous diagnosis of a serious mental health condition or psychiatric disorder
* Previous diagnosis of opioid use disorder or treatment for any substance use disorder
* Previously advised that yoga or massage is unsafe for their condition
* Current opioid use
* Current physical activity restrictions
* Planned surgery or procedures within 6 months of recruitment
* Planned travel outside the United States within treatment period time-frame
* Weight greater than or equal to 500 lbs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Mean System Usability Score | Assessed once after the results report has been sent to the participant, within 8 weeks of intervention completion
  Usability of the Personalized Trials platform will be evaluated using the System Usability Scale (SUS), a 10-item questionnaire created by Digital Equipment Co Ltd. and John Brooke in 1986 that asks users to score each item on a Likert scale from Strongly Disagree (1) to Strongly Agree (5). Individual results are calculated to arrive at a composite measure out of 100. Participant SUS scores will be averaged together. Higher scored values correlate to a more usable system, and therefore a better outcome.

SECONDARY OUTCOMES:
Mean Participant Satisfaction with Personalized Trials Components | Assessed once after the results report has been sent to the participant, within 8 weeks of intervention completion
  Participant satisfaction rated on a 5-point Likert scale from Very Dissatisfied (1) to Very Satisfied (5), or Strongly Disagree (1) to Strongly Agree (5). Higher scores correlate to greater satisfaction, and therefore a better outcome.
Mean Within-Subject Difference in Self-Reported Daily Pain Intensity During 3 Treatment Periods from Mean Baseline | From 2-Week Treatment Period 1 to 2-week Treatment Period 6
  Pain intensity is measured using the PROMIS Scale v1.0 - Pain Intensity 3a Fixed Length Short Form. The measure is modified from instructions to recall over the last 7 days to recall over the last 24 hours. Raw scores will be converted to an item response theory-based T-score using the PROMIS scoring manual. A T-score of 50 is the average for the US general population with an SD of 10. A higher T-score represents higher pain intensity or interference.
Mean Within-Subject Difference in Self-Reported Daily Pain Interference During 3 Treatment Periods from Mean Baseline | From 2-Week Treatment Period 1 to 2-week Treatment Period 6
  Pain interference is measured using a PROMIS Short Form v1.0 - Pain Interference 4a Fixed Length Short Form. The measure is modified from instructions to recall over the last 7 days to recall over the last 24 hours. Raw scores will be converted to an item response theory-based T-score using the PROMIS scoring manual. A T-score of 50 is the average for the US general population with an SD of 10. A higher T-score represents higher pain intensity or interference.
Mean Within-Subject Difference in Ecological Momentary Assessment Three-Times-Daily of Pain During 3 Treatment Periods from Mean Baseline | From 2-Week Treatment Period 1 to 2-week Treatment Period 6
  Numeric Pain Rating Scale adapted from McCaffery, Beebe et al. 1989 Numeric Pain Rating Scale, assessing current Pain level on a scale from 0 (none) to 10 (severe). Higher scores correlate to a worse outcome.
Mean Within-Subject Difference in Ecological Momentary Assessment Three-Times-Daily of Fatigue During 3 Treatment Periods from Mean Baseline | From 2-Week Treatment Period 1 to 2-week Treatment Period 6
  Numeric Fatigue Rating Scale adapted from McCaffery, Beebe et al. 1989, assessing current Fatigue level on a scale from 0 (none) to 10 (severe). Higher scores correlate to a worse outcome.
Mean Within-Subject Difference in Ecological Momentary Assessment Three-Times-Daily of Stress During 3 Treatment Periods from Mean Baseline | From 2-Week Treatment Period 1 to 2-week Treatment Period 6
  Numeric Stress Rating Scale adapted from McCaffery, Beebe et al. 1989, assessing current Stress level on a scale from 0 (none) to 10 (severe). Higher scores correlate to a worse outcome.
Mean Within-Subject Difference in Self-Reported Use of Pain Medication from Baseline | From 2-Week Treatment Period 1 to 2-week Treatment Period 6
  Average number of pain medication pills self-reported by participants as taken to manage their back pain. Daily question to quantify how many pain pills taken in the last 24 hours, and of what type and dosage.
Mean Within-Subject Difference in Device-Recorded Daily Steps from Mean Baseline | From 2-Week Treatment Period 1 to 2-week Treatment Period 6. Data collection to end after these 12 weeks.
  Average participant daily step data, as recorded by a Fitbit Charge 3 device.
Mean Within-Subject Difference in Device-Recorded Nightly Sleep from Mean Baseline | From 2-Week Treatment Period 1 to 2-week Treatment Period 6. Data collection to end after these 12 weeks.
  Average participant sleep minutes and sleep stage minute estimates, as recorded by a Fitbit Charge 3 device.

CONTACTS AND LOCATIONS:
Overall Officials: Karina W Davidson, PhD, MASc, Principal Investigator — Northwell Health
Locations (1):
- Center for Personalized Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) will be de-identified and pooled before sharing on the Open Science Framework, along with a data dictionary. Pooling N-of-1 trials together is a more efficient approach to deriving population-level estimates than conventional randomized controlled trials.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol, including the statistical analysis plan, will be made available in addition to the informed consent form before the first participant is randomized into the study. De-identified, pooled individual participant data will be made available within a year of final participant data collection. We anticipate this data to be available on the Open Science Framework platform indefinitely.
Access Criteria: All data and supporting information will be stored on the Open Science Framework, a free web application with no access restrictions.
URL: https://osf.io/ksfe6/